CLINICAL TRIAL: NCT05043103
Title: ELEGANCE - A Non-interventional Study on Long-term Effectiveness and Safety of Levodopa-Entacapone-Carbidopa Intestinal Gel (Lecigon®) in Patients With Advanced Parkinson's Disease in Routine Care
Brief Title: Long-Term Observational Study on Effectiveness and Safety of Lecigon in Patients With Advanced Parkinson's Disease
Acronym: ELEGANCE
Status: Active, not recruiting | Type: Observational
Sponsor: Britannia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-MA-2020-02
Record Dates: First submitted 2021-07-29; First posted 2021-09-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Parkinson Disease
Keywords: Parkinson´s Disease; Movement Disorders; Levodopa; Entacapone; Carbidopa Levodopa drug combination; Antiparkinson Agents; Anti-Dyskinesia-Agents; Dopamine Agents; Dopamine Agonists; Catechol-O-methyltransferase (COMT) inhibitor; Portable Pump; Gel; Quality of Life
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Lecigon® based on European Medicines Agency (EMA) SmPC — There might be different brand names in other countries

SUMMARY:
This observational study is designed to collect data on the use of the drug Lecigon® in daily clinical practice. The study is organised and funded by a pharmaceutical company called Britannia Pharmaceuticals Ltd (Britannia).

Lecigon® is prescribed by physicians in advanced Parkinson's disease when patients suffer from uncontrollable fluctuations in mobility, so-called motor fluctuations, which cannot be adjusted well with oral treatment, i.e. medication for swallowing.

In this study, data on the effect and possible side effects from everyday treatment with Lecigon® will be collected and scientifically evaluated. The study is intended to supplement the results of previous clinical studies with clinical data in routine medical care, collected from approximately 300 patients.

DETAILED DESCRIPTION:
Study design:

Non-interventional study, primary data collection.

No visits or measurements will be made mandatory by the observational plan. The assignment of patients to Lecigon® not decided in advance by the study's observational plan but falls within current practice. Prescription of Lecigon® occurred before and independently of the decision to include the patient in the study.

The participating centres will offer participation in the ELEGANCE study to all patients who receive treatment with Lecigon® part of routine clinical practice. From patients, who switched to treatment with Lecigon® prior to signing of informed consent, baseline data will be collected retrospectively.

The planned non-interventional study aims to collect real-world data on the effectiveness and safety of Lecigon® as a therapy for advanced Parkinson´s Disease in routine care in Germany and Austria. The study will be expanded to additional European countries as soon as marketing authorisation in these countries and commercial stock will be available.

Primary Objectives:

* Long-term effectiveness of Lecigon®
* Long-term safety of Lecigon®

Secondary Objectives:

* Patient non-motor symptoms and quality of life
* Healthcare resource utilisation by patients

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (18 years old and over) with Advanced Parkinson Disease already under treatment with Lecigon® (for up to 3 months before giving informed consent) in accordance with the Summary of Product Characteristics (SmPC)
* Patients or legal representative must have signed informed consent to participate in the study
* Patients are not taking part in another clinical (interventional) study at the same time

Exclusion Criteria:

* Patients with contraindications as defined in the current version of the SmPC for Lecigon®
* Patients who will not be seen again for their follow up care at the investigator's site after commencement of Lecigon® therapy
* Patients with pump placement or pump use issues, e.g. patients with acute severe illness, patients unable to perform pump therapy, and in case of lacking compliance due to severe dementia, agitation or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treating physician's normal patient pool
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in OFF time from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the effectiveness of Lecigon® treatment on the change in OFF time (h/day) from baseline up to 24 months, or treatment or study discontinuation as measured by Movement Disorder Society-Unified Parkinson's Disease Rating Scale IV Scores (MDS-UPDRS IV- motor complications)
Change in activities of daily living from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the effectiveness of Lecigon® treatment on the change in motor experiences of daily living from baseline up to 24 months, or treatment or study discontinuation as measured by Movement Disorder Society-Unified Parkinson's Disease Rating Scale II Scores (MDS-UPDRS II - motor experiences of daily living)
Change in Daily Levodopa dose from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the effectiveness of Lecigon® treatment on the change in Daily Levodopa dose [mg/day] from baseline up to 24 months, or treatment or study discontinuation as measured by morning bolus, continuous flow, extra boli, oral doses
Usage of other Anti-Parkinsonian medicinal products from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the effectiveness of Lecigon® treatment as measured by usage of other anti-Parkinsonian medicinal products (e.g. levodopa, dopamine agonists, Monoamine Oxidase (MAO)-B inhibitors, amantadine from baseline up to 24 months, or treatment or study discontinuation
Usage of the Lecigon® pump from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the effectiveness of Lecigon® treatment use of programmed pump rate (2 or 3 rates) from baseline up to 24 months, or treatment or study discontinuation will be collected
Change in Clinical Global Impression of Improvement (CGI-I) from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the effectiveness of Lecigon® treatment on the change in Clinical Global Impression of Improvement (CGI-I) from baseline up to 24 months, or treatment or study discontinuation as measured by Clinical Global Impression of Improvement Scale Score (CGI-I)
Change in Patient Global Impression of Change from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the effectiveness of Lecigon® treatment on the change in Patient Global Impression of Change (PGI-C) from baseline up to 24 months, or treatment or study discontinuation as measured by Patient Global Impression of Change Scale Score (PGI-C)
Satisfaction with treatment from baseline up to 24 months or treatment or study discontinuation | 24 months
  To assess the effectiveness with Lecigon®, satisfaction with treatment will be assessed in terms of pump size, weight, noise, handling and overall pump satisfaction from baseline up to 24 months or treatment or study discontinuation as measured by device satisfaction scale score between 0 (absolutely unsatisfied) to 10 (absolutely satisfied) for each item.
Occurrence of AEs and SAEs from baseline up to 24 months or treatment or study discontinuation | 24 months
  To assess the long-term safety of Lecigon® treatment Adverse Events (AEs) and Serious Adverse Events (SAEs) (including drug-related, device- and procedure-related Adverse Drug Reactions (ADRs) and Serious Adverse Drug Reactions (SADRs), AEs of special interest) from time of Informed consent to study completion for up to 24 months or treatment or study discontinuation will be collected

SECONDARY OUTCOMES:
Change in Non-Motor Symptoms from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on the change in Non-Motor Symptoms from baseline up to 24 months, or treatment or study discontinuation as measured by Non-Motor Symptom Scale Scores (NMSS)
Change in Sleep Quality from baseline up to 24 months, or treatment or study Discontinuation | 24 months
  To assess the impact of Lecigon® treatment on the change in sleep quality from baseline up to 24 months, or treatment or study discontinuation as measured by Parkinson's disease sleep Scale-2 Score (PDSS-2)
Change in Activities of daily living from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on the change in activities of daily living from baseline up to 24 months, or treatment or study discontinuation as measured by Movement Disorder Society-Unified Parkinson's Disease Rating Scale Ib Score (MDS-UPDRS Ib - non-motor experiences of daily living)
Change in Quality of Life from baseline up to 24 months or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on the change in quality of life from baseline up to 24 months, or treatment or study discontinuation as measured by Parkinson's Disease Questionnaire total score (PDQ-8 or PDQ-39)
Usage of Healthcare resources from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on usage of Healthcare resources as measured by additional hospitalisation due to complications out of scope of nurse support team since the last visit

OTHER OUTCOMES:
Change in Body weight from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on vital signs as measured by change in the Body weight (Kg) from baseline up to 24 months, or treatment or study discontinuation
Change in Blood pressure from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on vital signs as measured by change in the Blood pressure (mmHg) from baseline up to 24 months, or treatment or study discontinuation
Change in Pulse from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on vital signs as measured by change in the Pulse (bpm) from baseline up to 24 months, or treatment or study discontinuation
Change in the Liver function tests from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on laboratory results as measured by change in the Liver function tests from baseline up to 24 months or treatment or study discontinuation
Change in the full blood count from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on laboratory results as measured by change in the full blood count including B12 metabolism panel from baseline up to 24 months or treatment or study discontinuation
Change in the ECG from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on laboratory results as measured by change in the ECG from baseline up to 24 months or treatment or study discontinuation
Change in the Renal function tests from baseline up to 24 months, or treatment or study discontinuation | 24 months
  To assess the impact of Lecigon® treatment on laboratory results as measured by change in the Renal function tests from baseline up to 24 months or treatment or study discontinuation

CONTACTS AND LOCATIONS:
Locations (56):
- Austria (4):
  - Universitätsklinik für Neurologie, Medizinische Universität Graz, Graz
  - Abteilung für Neurologische Rehabilitation, Gailtal-Klinik, Hermagor
  - Universitätsklinik für Neurologie, Medizinische Universität Innsbruck, Innsbruck
  - Kepler Universitätsklinikum, Linz
- Belgium (5):
  - AZ Sint-Jan, Bruges
  - Antwerp University Hospital, Edegem
  - Ghent University Hospital, Ghent
  - University Hospital Liege, Liège
  - Centre Hospitalier de Wallonie picarde (Chwapi), Tournai
- Sveti Naum, Sofia, Bulgaria
- Croatia (4):
  - UHC Osijek, J. Klinici za neurologiju, Osijek
  - University Hospital Centre Rijeka (KBC Rijeka), Rijeka
  - Klinička bolnica Dubrava, Zagreb
  - University Hospital Centre (KBC Zagreb), Zagreb
- Czechia (2):
  - Masaryk university, Brno
  - Fakultní nemocnice Olomouc, Olomouc
- Bispebjerg Hospital, Copenhagen, Denmark
- Germany (13):
  - Segeberger Kliniken GmbH Neurologisches Zentrum, Bad Segeberg
  - Kliniken Beelitz GmbH Neurologisches Fachkrankenhaus für Bewegungsstörungen/Parkinson, Beelitz-Heilstätten
  - Charité - Universitätsmedizin Berlin, Berlin
  - Uniklinik Köln, Cologne
  - Krankenhaus Lindenbrunn, Coppenbrügge
  - Klinik für Neurologie - Universitätsklinikum Essen, Essen
  - Zentrum für Seltene Erkrankungen Göttingen, Göttingen
  - Universitätsklinikum Giessen und Marburg, Marburg
  - Evangelisches Krankenhaus Oldenburg, Oldenburg
  - Klinikum Osnabrück GmbH Klinik für Neurologie, Osnabrück
  - Universitätsklinikum Tübingen, Tübingen
  - RKU - Universitäts und Rehabilitationskliniken Ulm gGmbH, Ulm
  - Parkinson-Klinik Ortenau, Wolfach
- Hungary (3):
  - Semmelweis Egyetem Neurológiai Klinika Budapest, Budapest
  - Pécsi Tudományegyetem Klinikai Központ Szemészeti Klinika, Pécs
  - SZTE Szent-Györgyi Albert Klinikai Közpon, Szeged
- Ireland (2):
  - St. Vincent's University Hospital, Dublin
  - The Dublin Neurological Institute, Mater Hospital, Dublin
- University Medical Center Groningen, Groningen, Netherlands
- Romania (10):
  - Emergency Hospital Brasov, Spitalul Clinic Județean de Urgență Brașov, Brasov
  - Spitalul Universitar de Urgență Elias, Bucharest
  - Colentina Hospital Bucharest, Bucharest
  - Bucharest University Emergency Hospital, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - County Emergency Hospital Cluj-Napoca, Cluj-Napoca
  - County Clinical Emergency Hospital of Constanta, Constanța
  - Emergency County Hospital Targu Mures, Târgu Mureş
  - Timiş County Emergency Clinical Hospital- Neurology 1, Timișoara
  - Timiş County Emergency Clinical Hospital, Timișoara
- Slovenia (2):
  - Department of Neurology, University Medical Centre, Ljubljana
  - Univerzitetni klinični center Maribor, Maribor
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital Virgen del Rocio, Seville
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skånes universitetssjukhus Lund, Lund
  - Uppsala university hospital, Uppsala